CLINICAL TRIAL: NCT00130923
Title: Risperidone Long-Acting for Alcohol and Schizophrenia Treatment (R-LAST)
Brief Title: Risperidone Long-acting Versus Oral Risperidone in Patients With Schizophrenia and Alcohol Use Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Alan Green, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17359; RIS-EMR-4032
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Results first posted 2012-10-24 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia; Psychotic Disorders; Substance Abuse; Alcohol Abuse
Keywords: Risperidone; Schizophrenia; Substance Use Disorder; Alcohol Use Disorder; Treatment; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Substance-Related Disorders; Alcoholism | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risperidone Long Acting (Experimental): Risperidone Long Acting; aka Risperdal Consta; injectable form
  Interventions: Drug: Risperidone Long Acting
- Oral Risperidone (Active Comparator): Oral Risperidone; aka Risperdal; oral form
  Interventions: Drug: oral risperidone

INTERVENTIONS:
Drug: Risperidone Long Acting — Dose 25.00, 37.50 or 50.00 mg q two weeks
  Other Names: Risperdal Consta
  Arms: Risperidone Long Acting
Drug: oral risperidone — 0.50-6.00 mg oral risperidone daily
  Other Names: Risperdal
  Arms: Oral Risperidone

SUMMARY:
The purpose of this study is to compare the efficacy of oral risperidone (Risperdal) to risperidone long-acting (Consta) in reducing alcohol use in persons diagnosed with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Comorbid alcohol/substance use disorder (SUD) in people with schizophrenia is a major concern, both in view of the high frequency of SUD among patients with schizophrenia and the difficulty in managing such patients. Though antipsychotic medications are effective in reducing symptoms and impairment in persons with schizophrenia, the typical antipsychotic agents are of limited value in controlling alcohol/substance use in these patients. Extrapyramidal, dysphoric side effects of conventional neuroleptics may actually promote the use of substances in an attempt to counteract these effects. In addition, medication non-compliance is common among patients with schizophrenia.

Novel antipsychotics have altered treatment expectations and outcomes for patients with severe forms of schizophrenia. A growing number of studies have assessed the effects of oral risperidone in persons with dual disorders. Potential mechanisms of action by which risperidone and other atypical antipsychotics could decrease substance use include being less likely to cause extrapyramidal side effects than typical agents, improving negative symptoms and ameliorating a dysfunction of the brain reward system. Risperidone long-acting injectable medication addresses issues of noncompliance, while avoiding peak blood levels of oral preparations, thereby minimizing EPS and improving negative symptoms of schizophrenia. Risperidone may also facilitate dopamine neurotransmission in the prefrontal cortex and correct a hypothesized dysfunction of the brain reward system.

This study is an open, randomized, controlled study to compare intramuscular long-acting risperidone to oral risperidone with blinded ratings to determine whether the long-acting form of risperidone has greater efficacy in reducing substance use. Patients with schizophrenia or schizoaffective disorder, age 18 to 65, who are taking any single oral antipsychotic medication except clozapine or risperidone long-acting may be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Schizophrenia or schizoaffective disorder
* Meets the Structured Clinical Interview for DSM-IV (SCID) criteria for an alcohol use disorder
* Alcohol use on at least 5 days during the 4 weeks prior to randomization
* Patient is medically stable to start either form of risperidone.

Exclusion Criteria:

* Current treatment with clozapine.
* Current treatment with injectable risperidone long-acting.
* Currently pregnant, planning to become pregnant, or unwilling to use an acceptable form of birth control.
* Change in medications (dose of current medication, discontinuation of medication, or new medication) in past 30 days.
* History of or current breast cancer.
* History of intolerance of or allergy to risperidone or risperidone long-acting.
* Currently residing in a residential program designed to treat substance use disorders.
* Current treatment with long-acting, injectable antipsychotic medication will require a review by the medication adjustment group before entering the client into the study.
* Past treatment with risperidone long-acting will require a review by the medication adjustment group before entering the client into the study.
* Treatment at baseline with a second antipsychotic medication will require a review by the medication adjustment group before entering the client into the study.
* Treatment at baseline with a psychotropic agent proposed to curtail substance use will require a review by the medication adjustment group before entering the client into the study.
* Patients who, in the opinion of the investigator, are judged unsuitable to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan I. Green, MD, Principal Investigator — Dartmouth Medical School, Dartmouth College
Locations (8):
- United States (8):
  - JMH Mental Health Center, University of Miami, Miami, Florida
  - School of Pharmacy, Univ. of Missouri Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - West Central Behavioral Health, Lebanon, New Hampshire
  - Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - Center for Psychiatric Advancement, Nashua, New Hampshire
  - University of South Carolina, Columbia, South Carolina
  - White River Junction Veterans Admininistration Medical Center, White River Junction, Vermont

REFERENCES:
- [Background] Albanese MJ, Khantzian EJ, Murphy SL, Green AI. Decreased substance use in chronically psychotic patients treated with clozapine. Am J Psychiatry. 1994 May;151(5):780-1. doi: 10.1176/ajp.151.5.780b. No abstract available. PMID 8166327
- [Background] Albanese M. Risperidone in substance abusers with bipolar disorder. Presented at the 39th Annual Meeting of the American College of Neuropsychopharmacology. Sa Juan, PR, 2000.
- [Background] Akaike, H, Information theory and an extension of the maximum likelihood principle., in 2nd International Symposium on Information Theory and Control., EBN Petrovand & C. Csaki, Editors. 1973, Akademia Kiado: Budapest, p. 267-281.
- [Background] Bartels SJ, Teague GB, Drake RE, Clark RE, Bush PW, Noordsy DL. Substance abuse in schizophrenia: service utilization and costs. J Nerv Ment Dis. 1993 Apr;181(4):227-32. doi: 10.1097/00005053-199304000-00003. PMID 8473874
- [Background] Birkett MA, Day SJ. Internal pilot studies for estimating sample size. Stat Med. 1994 Dec 15-30;13(23-24):2455-63. doi: 10.1002/sim.4780132309. PMID 7701146
- [Background] Bowers MB Jr, Mazure CM, Nelson JC, Jatlow PI. Psychotogenic drug use and neuroleptic response. Schizophr Bull. 1990;16(1):81-5. doi: 10.1093/schbul/16.1.81. PMID 1970670
- [Background] Buckley P, Thompson P, Way L, Meltzer HY. Substance abuse among patients with treatment-resistant schizophrenia: characteristics and implications for clozapine therapy. Am J Psychiatry. 1994 Mar;151(3):385-9. doi: 10.1176/ajp.151.3.385. PMID 8109646
- [Background] Buckley P, Thompson PA, Way L, Meltzer HY. Substance abuse and clozapine treatment. J Clin Psychiatry. 1994 Sep;55 Suppl B:114-6. PMID 7961553
- [Background] Buckley PF. Novel antipsychotic medications and the treatment of comorbid substance abuse in schizophrenia. J Subst Abuse Treat. 1998 Mar-Apr;15(2):113-6. doi: 10.1016/s0740-5472(97)00134-7. PMID 9561949
- [Background] Buckley PF. Substance abuse in schizophrenia: a review. J Clin Psychiatry. 1998;59 Suppl 3:26-30. PMID 9541335
- [Background] Buckley PF, Miller A, Chiles JA, Sajatovic M. Implementing effectiveness research and improving care for schizophrenia in real-world settings. Am J Manag Care. 1999 Jun 25;5 Spec No:SP47-56. PMID 10538860
- [Background] Buckley P, McCarthy M, Chapman P, Richman C, Yamamoto B. Clozapine treatment of comorbid substance abuse in patients with schizophrenia. Schizophr Res 1999, 36:272.
- [Background] Coldham EL, Addington J, Addington D. Medication adherence of individuals with a first episode of psychosis. Acta Psychiatr Scand. 2002 Oct;106(4):286-90. doi: 10.1034/j.1600-0447.2002.02437.x. PMID 12225495
- [Background] Drake RE, Xie H, McHugo GJ, Green AI. The effects of clozapine on alcohol and drug use disorders among patients with schizophrenia. Schizophr Bull. 2000;26(2):441-9. doi: 10.1093/oxfordjournals.schbul.a033464. PMID 10885642
- [Background] Frison L, Pocock SJ. Repeated measures in clinical trials: analysis using mean summary statistics and its implications for design. Stat Med. 1992 Sep 30;11(13):1685-704. doi: 10.1002/sim.4780111304. PMID 1485053
- [Background] Green AI, Zimmet SV, Strous RD, Schildkraut JJ. Clozapine for comorbid substance use disorder and schizophrenia: do patients with schizophrenia have a reward-deficiency syndrome that can be ameliorated by clozapine? Harv Rev Psychiatry. 1999 Mar-Apr;6(6):287-96. doi: 10.3109/10673229909017206. PMID 10370435
- [Background] Green AI, Salomon MS, Brenner MJ, Rawlins K. Treatment of schizophrenia and comorbid substance use disorder. Curr Drug Targets CNS Neurol Disord. 2002 Apr;1(2):129-39. doi: 10.2174/1568007024606230. PMID 12769622
- [Background] Green AI, Burgess ES, Dawson R, Zimmet SV, Strous RD. Alcohol and cannabis use in schizophrenia: effects of clozapine vs. risperidone. Schizophr Res. 2003 Mar 1;60(1):81-5. doi: 10.1016/s0920-9964(02)00231-1. PMID 12505141
- [Background] Hunt GE, Bergen J, Bashir M. Medication compliance and comorbid substance abuse in schizophrenia: impact on community survival 4 years after a relapse. Schizophr Res. 2002 Apr 1;54(3):253-64. doi: 10.1016/s0920-9964(01)00261-4. PMID 11950550
- [Background] Khantzian EJ. The self-medication hypothesis of addictive disorders: focus on heroin and cocaine dependence. Am J Psychiatry. 1985 Nov;142(11):1259-64. doi: 10.1176/ajp.142.11.1259. PMID 3904487
- [Background] Khantzian EJ. The self-medication hypothesis of substance use disorders: a reconsideration and recent applications. Harv Rev Psychiatry. 1997 Jan-Feb;4(5):231-44. doi: 10.3109/10673229709030550. PMID 9385000
- [Background] Lacro JP, Dunn LB, Dolder CR, Leckband SG, Jeste DV. Prevalence of and risk factors for medication nonadherence in patients with schizophrenia: a comprehensive review of recent literature. J Clin Psychiatry. 2002 Oct;63(10):892-909. doi: 10.4088/jcp.v63n1007. PMID 12416599
- [Background] Laird NM, Ware JH. Random-effects models for longitudinal data. Biometrics. 1982 Dec;38(4):963-74. PMID 7168798
- [Background] Lee, ET. Statistical Methods for Survival Analysis. 1992, New York: John Wiley & Sons.
- [Background] Newton TF, Ling W, Kalechstein AD, Uslaner J, Tervo K. Risperidone pre-treatment reduces the euphoric effects of experimentally administered cocaine. Psychiatry Res. 2001 Jul 24;102(3):227-33. doi: 10.1016/s0165-1781(01)00255-4. PMID 11440773
- [Background] Salyers MP, Mueser KT. Social functioning, psychopathology, and medication side effects in relation to substance use and abuse in schizophrenia. Schizophr Res. 2001 Mar 1;48(1):109-23. doi: 10.1016/s0920-9964(00)00063-3. PMID 11278158
- [Background] Siris SG. Pharmacological treatment of substance-abusing schizophrenic patients. Schizophr Bull. 1990;16(1):111-22. doi: 10.1093/schbul/16.1.111. PMID 1970669
- [Background] Smelson DA, Losonczy MF, Davis CW, Kaune M, Williams J, Ziedonis D. Risperidone decreases craving and relapses in individuals with schizophrenia and cocaine dependence. Can J Psychiatry. 2002 Sep;47(7):671-5. doi: 10.1177/070674370204700710. PMID 12355680
- [Background] Tukey, JW. Exploratory Data Analysis. 1977, Reading, MA: Addison Wesley Publ. Co.
- [Background] Waternaux, C, Laird, N, Ware, J. Methods for the analysis of longitudinal data: Blood concentrations and cognitive development. J.Amer. Stat. Assoc. 1989: 84, p.33-41.
- [Background] Weiss RE, Lazaro CG. Residual plots for repeated measures. Stat Med. 1992 Jan 15;11(1):115-24. doi: 10.1002/sim.4780110110. PMID 1557567
- [Background] Zimmet SV, Strous RD, Burgess ES, Kohnstamm S, Green AI. Effects of clozapine on substance use in patients with schizophrenia and schizoaffective disorder: a retrospective survey. J Clin Psychopharmacol. 2000 Feb;20(1):94-8. doi: 10.1097/00004714-200002000-00016. PMID 10653215
- [Derived] Green AI, Brunette MF, Dawson R, Buckley P, Wallace AE, Hafez H, Herz M, Narasimhan M, Noordsy DL, O'Keefe C, Sommi RW, Steinbook RM, Weeks M. Long-acting injectable vs oral risperidone for schizophrenia and co-occurring alcohol use disorder: a randomized trial. J Clin Psychiatry. 2015 Oct;76(10):1359-65. doi: 10.4088/JCP.13m08838. PMID 26302441

RESULTS

PARTICIPANT FLOW:
Groups:
- Risperidone Long Acting Injectable (LAI): Risperidone Long Acting Injectable (LAI), begun with 25 mg dose given intramuscularly(IM)every two weeks. The dose was titrated up to a target dose of 37.5 mg IM, with injections given every two weeks. The maximum dose of LAI risperidone was 50 mg every two weeks.
- Oral Risperidone Aka Risperdal: Oral Risperidone aka Risperdal. Participants who were randomized to take oral risperidone were titrated over two weeks up to a target dose of 4 mg per day. The maximum daily dose of oral risperidone was 6 mg.
Period: Overall Study
Arm/Group | Risperidone Long Acting Injectable (LAI) | Oral Risperidone Aka Risperdal
Started | 49 | 46
Completed | 36 | 32
Not Completed | 13 | 14

BASELINE CHARACTERISTICS:
Groups:
- Oral Risperidone Aka Risperal: Oral Risperidone aka Risperdal. Participants who were randomized to take oral risperidone were titrated over two weeks up to a target dose of 4 mg per day. The maximum daily dose of oral risperidone was 6 mg.
- Total: Total of all reporting groups
Arm/Group | Risperidone Long Acting Injectable (LAI) | Oral Risperidone Aka Risperal | Total
Number analyzed (Participants) | 49 | 46 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 46 | 95
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (10.1) | 41.7 (11.5) | 41.70 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 37 | 36 | 73
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 46 | 95

OUTCOME MEASURES:

1. Primary Outcome: Change Over Time in Frequency of Heavy Drinking Days (Used to Evaluate Treatment Efficacy)
Description: Frequency of heavy drinking days is obtained each week retrospectively as the number of heavy drinking days during the prior week (assessed by the Timeline Followback Scale). A heavy drinking day is defined as 4 or more drinks per day for a female and 5 or more drinks per day for a male. Mixed models are used to obtain estimates of efficacy from the partial data provided by each subject while adherent to assigned treatment (under the 'missing at random' assumption). The 'explanatory' estimands (target of the mixed model estimation) are defined in terms of population quantities that would have occurred had all subjects remained on assigned treatment throughout the study. The point estimate for each arm is reported under Number.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: heavy drinking days per week
Arm/Group | Risperidone Long Acting Injectable (LAI) | Oral Risperidone Aka Risperal
Number analyzed (Participants) | 49 | 46
heavy drinking days per week | -.11 [-1.12 to .9] | .68 [.083 to 1.28]
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectable (LAI) vs Oral Risperidone Aka Risperal; Test type: Superiority; p = 0.054, Mixed Models Analysis; difference in treatment slopes = -.043, Standard Error of Mean .021 — We report the estimated coefficient for difference in treatment slopes in a mixed model and its standard error

2. Secondary Outcome: Average Over Time of Frequency of Drinking Days (Used to Evaluate Treatment Efficacy)
Description: Frequency of drinking days is obtained each week retrospectively as the number of drinking days during the prior week (assessed using the Timeline Followback). Mixed models are used to obtain estimates of efficacy from the partial data provided by each subject while adherent to assigned treatment (under the 'missing at random' assumption). The 'explanatory' estimands (target of the mixed model estimation) are defined in terms of population quantities that would have occurred had all subjects remained on assigned treatment throughout the study. The point estimate for each arm is reported under Number.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: drinking days per week
Arm/Group | Risperidone Long Acting Injectable (LAI) | Oral Risperidone Aka Risperdal
Number analyzed (Participants) | 49 | 46
drinking days per week | 2.84 [1.72 to 3.95] | 3.46 [2.5 to 4.42]
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectable (LAI) vs Oral Risperidone Aka Risperdal; Test type: Superiority; p = .035, Mixed Models Analysis; Difference in treatment means = -.62, Standard Error of Mean .29 — We report the estimated coefficient for difference in treatment means in a mixed model and its standard error

3. Secondary Outcome: Average Over Time of Severity of Illness and Global Improvement (Used to Evaluate Treatment Efficacy)
Description: A rater assesses the severity of illness and global impression using a scale from 1 to 7 (Clinical Global Impression), where higher values represent a worse outcome. Mixed models are used to obtain estimates of efficacy from the partial data provided by each subject while adherent to assigned treatment (under the 'missing at random' assumption). The 'explanatory' estimands (target of the mixed model estimation) are defined in terms of population quantities that would have occurred had all subjects remained on assigned treatment throughout the study. The point estimate for each arm is reported under Number.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: ordinal unit of severity
Arm/Group | Risperidone Long Acting Injectable (LAI) | Oral Risperidone Aka Risperal
Number analyzed (Participants) | 49 | 46
ordinal unit of severity | 4.02 [3.13 to 4.91] | 3.96 [3.08 to 4.83]
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectable (LAI) vs Oral Risperidone Aka Risperal; Test type: Superiority; p = .57, Mixed Models Analysis; difference in treatment means = .056, Standard Error of Mean .099 — We report the estimated coefficient for difference in treatment means in a mixed model and its standard error

4. Secondary Outcome: Average Over Time of Positive and Negative Symptoms (Used to Evaluate Treatment Efficacy)
Description: A rater assesses positive and negative symptoms of schizophrenia using a 30-item scale (Positive and Negative Symptom Score) Scores range from 30 to 210, where higher values represent a worse outcome. Mixed models are used to obtain estimates of efficacy from the partial data provided by each subject while adherent to assigned treatment (under the 'missing at random' assumption). The 'explanatory' estimands (target of the mixed model estimation) are defined in terms of population quantities that would have occurred had all subjects remained on assigned treatment throughout the study. The point estimate for each arm is reported under Number.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: ordinal severity of symptoms
Arm/Group | Risperidone Long Acting Injectable (LAI) | Oral Risperidone Aka Risperdal
Number analyzed (Participants) | 49 | 46
ordinal severity of symptoms | 78.2 [64.9 to 91.5] | 75.5 [65.3 to 89.7]
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectable (LAI) vs Oral Risperidone Aka Risperdal; Test type: Superiority; p = .32, Mixed Models Analysis; difference in treatment means = 2.65, Standard Error of Mean 2.68 — We report the estimated coefficient difference in treatment means in a mixed model and its standard error

5. Secondary Outcome: Average Over Time of Global Functioning (Used to Evaluate Treatment Efficacy)
Description: A rater assesses social, occupational and psychological functioning on a hypothetical continuum of mental health - illness (using Global Assessment of Functioning); scores range from 100 to 1, where higher values represent a better outcome. Mixed models are used to obtain estimates of efficacy from the partial data provided by each subject while adherent to assigned treatment (under the 'missing at random' assumption). The 'explanatory' estimands (target of the mixed model estimation) are defined in terms of population quantities that would have occurred had all subjects remained on assigned treatment throughout the study. The point estimate for each arm is reported under Number.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: ordinal severity of impairment
Arm/Group | Risperidone Long Acting Injectable (LAI) | Oral Risperidone Aka Risperdal
Number analyzed (Participants) | 49 | 46
ordinal severity of impairment | 50.8 [42.7 to 58.9] | 49.9 [42.2 to 57.6]
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectable (LAI) vs Oral Risperidone Aka Risperdal; Test type: Superiority; p = .44, Mixed Models Analysis; difference in treatment means = .93, Standard Error of Mean 1.19 — We report the estimated coefficient for difference in treatment means in a mixed model and its standard error

6. Secondary Outcome: Number of Participants With Medication Adherence
Description: Number of participants with medication adherence (defined as taking medication at least 75% of the days in the treatment period).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Risperidone Long Acting Injectable (LAI) | Oral Risperidone Aka Risperdal
Number analyzed (Participants) | 49 | 46
Participants | 43 | 28
Statistical Analysis 1: Comparison: Risperidone Long Acting Injectable (LAI) vs Oral Risperidone Aka Risperdal; Test type: Superiority; p = .003, Chi-squared; Statistical test of hypothesis. Value of the Chi-squared statistic is 9.08

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Risperidone Long Acting Injectable (LAI) | Oral Risperidone Aka Risperal
Serious Adverse Events (participants affected / at risk) | 16/49 | 12/46
Other Adverse Events (participants affected / at risk) | 27/49 | 14/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone Long Acting Injectable (LAI) (N=49) | Oral Risperidone Aka Risperal (N=46)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Delerium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 1 (1)
Epitaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Injury, poisongin and procedural complications - Other, specify - Gunshot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Psychiatric Disorders - Other, specify - unspecified (Psychiatric disorders) | 1 (1) | 1 (1)
Psychiatric Disorders - Other, specify Substance Dependence (Psychiatric disorders) | 2 (2) | 1 (8)
Psychosis (Psychiatric disorders) | 2 (2) | 5 (6)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 2 (5)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risperidone Long Acting Injectable (LAI) (N=49) | Oral Risperidone Aka Risperal (N=46)
Anxiety (Psychiatric disorders) | 4 (4) | 1 (1)
Depression (Psychiatric disorders) | 4 (6) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 2 (2)
Erectile Disfunction (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Gastrointestinal Disorder - Other, Hypersalivation (Gastrointestinal disorders) | 3 (4) | 0 (0)
Injection Site Reactions (General disorders) | 3 (15) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (8) | 3 (3)
Musculo-Skeletal Connective Tissue Disorder-Other, Muscle Stiffness (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0)
Pain (General disorders) | 5 (5) | 0 (0)
Psychiatric Disorders - Other, Specify: Substance Dependence (Psychiatric disorders) | 1 (2) | 3 (5)
Somnolence (Nervous system disorders) | 4 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No